CLINICAL TRIAL: NCT00061737
Title: Quality of Life in Pediatric Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: QLPIMB (completed)
Record Dates: First submitted 2003-06-03; First posted 2003-06-04 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Pediatric IBD; Inflammatory; Bowel
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Measurement of the quality of life (QoL) of children and adolescents with inflammatory bowel diseases (IBD) has had little attention, despite the importance of understanding key factors affecting QoL, especially for measuring the effects of clinical trials to improve IBD outcomes. The main purpose of this pilot study is to examine the impact of clinical severity and treatment social factors on the quality of life (QoL) of a diverse population of children and adolescents with inflammatory bowel disease (IBD). Secondary purposes include determining the effects of sociodemographic factors on QoL and exploring the concordance of views of parents and children of QoL. The study aims are to 1) determine the associations of of clinical characteristics (condition type, activity/severity, and treatment) with specific components of general health-related quality of life and IBD-specific QoL; 2) describe the effects of sociodemographic characteristics (SES, age, and gender) on these measures; and 3) compare the views of different observers (parent and child with IBD) of the child's QoL. The study will apply both general and condition-specific QoL measures among a random sample of 250 children and adolescents with IBD, ages 5-18 years, in six clinical sites. We will obtain measures of QoL from both the child and a parent in each case. The study will obtain additional data regarding the subjects' clinical condition (condition type, severity/activity, treatment [including surgery], age of onset) and socioeconomic status (household structure and income). Main analyses will compare general and specific measures of QoL and examine the influence of clinical and sociodemographic variables on QoL, through multivariate regression techniques. We will also examine the differences in child and parent assessments of QoL. The information from this study will provide a stronger base for future studies of treatment and natural history of IBD. It will help to clarify the life domains that are affected by IBD and will inform interventions to improve QoL for children with IBD.

ELIGIBILITY:
All children ages 8-17 years in any of six centers for inflammatory bowel disease in children who have already enrolled in the IBD consortium database.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 350 (Estimated)
Dates: Start 2003-01

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California San Francisco, San Francisco, California
  - Children's Health Care of Atlanta, Atlanta, Georgia
  - University of Chicago Children's Hospital, Chicago, Illinois
  - MassGeneral Hospital for Children, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas